CLINICAL TRIAL: NCT04091659
Title: Use of Virtual Reality for Overdose Management Educational Trainings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Nicholas Giordano, PhD, RN, Lecturer, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 833978
Record Dates: First submitted 2019-09-11; First posted 2019-09-17 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Drug Overdose; Virtual Reality
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Education (Active Comparator): Standard Educational (Control): The public health department's training includes printed handouts on how to administer naloxone and youtube videos on how to spot signs and symptoms of overdose and administer naloxone. Additionally, staff are on hand to provide one on one verbal educational trainings to local community members voluntarily seeking education.
  Interventions: Other: Standard Education
- Virtual Reality (Experimental): Virtual Reality Education (Intervention): The experimental group of libraries will receive the virtual reality simulation, which is guided by the NLN Jeffries Simulation Theory, and lasts 9 minutes. The virtual reality education is based on scenes and dialogue conducted during the hybrid high-fidelity simulation, from a script developed using the existing hybrid simulation on opioid overdose intervention. This virtual reality education is an educational intervention.
  Interventions: Other: Virtual Reality Education

INTERVENTIONS:
Other: Virtual Reality Education — Virtual Reality Education (Intervention): The experimental group of libraries will receive the virtual reality simulation, which is guided by the NLN Jeffries Simulation Theory, and lasts 9 minutes. The virtual reality education is based on scenes and dialogue conducted during the hybrid high-fidelity simulation, from a script developed using the existing hybrid simulation on opioid overdose intervention. This virtual reality education is an educational intervention.
  Arms: Virtual Reality
Other: Standard Education — Standard Educational (Control): The public health department's training includes printed handouts on how to administer naloxone and youtube videos on how to spot signs and symptoms of overdose and administer naloxone. Additionally, staff are on hand to provide one on one verbal educational trainings to local community members voluntarily seeking education.
  Arms: Standard Education

SUMMARY:
This cluster-randomized trial will compare changes in attitudes and knowledge on administering naloxone based on exposure to either a virtual reality educational training or the current standard educational trainings (e.g. on-line videos, printed information handouts) offered at local libraries. Individuals attending local library's naloxone training days will voluntarily complete an anonymous validated survey pre and post attending either the virtual reality or standard educational training.

DETAILED DESCRIPTION:
This study will utilize a cluster-randomized trial design. Entire libraries will be randomized to either offer community members the virtual reality training or the standard educational offerings (e.g. handouts, online videos). Volunteers will be asked to complete the brief, anonymous, and validated Opioid Overdose Knowledge Scale prior to receiving an education intervention (pretest) and then again immediately after (posttest). Neither participants nor investigators will be blinded. Library patrons who do not participate in the study will be offered current standard training materials. Regardless of the library's randomization, to either virtual reality or standard training, all patrons completing pre and post test surveys will have the opportunity to view the virtual reality training or other public health department materials.

ELIGIBILITY:
Inclusion Criteria:

* Able to complete paper surveys independently
* Provide verbal consent

Exclusion Criteria:

* Unable to complete immediate post-training assessment
* Individuals under 18 years of age
* Individuals who cannot communicate in English and provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Giordano, Principal Investigator — Lecturer
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be made available upon request with approved IRB from requesting institution
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after study completion and up to 3 years later
Access Criteria: Made available upon request and with approved IRB from requesting institution

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Education | Virtual Reality
Started | 40 | 58
Completed | 37 | 57
Not Completed | 3 | 1
Not completed — Protocol Violation | 3 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Education | Virtual Reality | Total
Number analyzed (Participants) | 37 | 57 | 94
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [25 to 55] | 41 [30 to 60] | 40 [27 to 57]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 12 | 22 | 34
  Female | 24 | 33 | 57
  Nonbinary | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 13 | 24
  White | 14 | 21 | 35
  More than one race | 12 | 23 | 35
  Unknown or Not Reported | 0 | 0 | 0
OOKS [Median (Inter-Quartile Range); unit: units on a scale] — Scores range from 0 to 10, with higher scores indicating greater knowledge on how to identify and appropriately intervene during an opioid related overdose, including proper use of naloxone", or similar
  units on a scale | 5 [4 to 6] | 5 [3 to 7] | 5 [4 to 6]
OOAS [Median (Inter-Quartile Range); unit: units on a scale] — OOAS items were scored on a Likert-type scale and higher scores suggested more favorable attitudes towards opioid overdose response, where 1=completely disagree, and 5=completely agree
  units on a scale | 3.3 [3.1 to 3.6] | 3.4 [3.0 to 3.9] | 3.4 [3.0 to 3.7]

OUTCOME MEASURES:

1. Primary Outcome: Change in Opioid Overdose Knowledge Scale (OOKS) From Pre- to Post-training
Description: Higher scores on the OOKS indicate greater knowledge on how to identify and appropriately intervene during an opioid related overdose, including proper use of naloxone. The tool has been validated with healthcare professionals and lay persons and used to assess changes in knowledge and attitudes after in-person naloxone trainings. This main outcome of this study is examining changes in the OOKS subscale for signs of an opioid overdose with scores ranging from 0 to 10.
Time Frame: Immediately Pre-Training and Within 1 Hour Post-training
Population: Higher difference in scores indicates greater improvement from baseline to follow up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Education | Virtual Reality
Number analyzed (Participants) | 37 | 57
units on a scale | 2 [1 to 2] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Standard Education vs Virtual Reality; Test type: Equivalence — To determine if the two training approaches were comparable to one another a margin of +/- 1 was used in differences of both OOKS and OOAS scale scores based on previously established literature. An equivalence test of differences using two one-sided tests on data from a cluster-randomized design was conducted using structural equation modeling. Sample sizes of 35 and 57 in group two, obtained by sampling 9 clusters, achieve 85% power to detect equivalence. The significance level is 0.05; p = 0.65, SEM; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.85 to 0.49]; The control group, standard education was the reference for this model

2. Secondary Outcome: Change in Opioid Overdose Attitudes Scale (OOAS) From Pre- to Post-training
Description: The OOAS subscales assessing competencies to manage an opioid overdose (5 items). Study participants were given intranasal naloxone, so all items were adapted to refer to intranasal naloxone rather than injectable naloxone. OOAS items were scored on a Likert-type scale and higher scores suggested more favorable attitudes towards opioid overdose response, where 1=completely disagree, and 5=completely agree
Time Frame: Immediately Pre-Training and Within 1 Hour Post-training
Population: Higher difference in scores indicates greater improvement from baseline to follow up
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Education | Virtual Reality
Number analyzed (Participants) | 37 | 57
units on a scale | 1 [0.57 to 4.9] | 1 [0.71 to 1.43]
Statistical Analysis 1: Comparison: Standard Education vs Virtual Reality; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.02, SEM; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.02 to 0.50] — The control group, standard education, was the reference

ADVERSE EVENTS:
Time Frame: Not monitored/assessed
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Standard Education | Virtual Reality
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT04091659/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT04091659/ICF_001.pdf